CLINICAL TRIAL: NCT06379477
Title: Correction of Refractive Error Surprises After Cataract Surgery in Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed saad, ophthalmology specialist at ophthalmology department Assiut University hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: refractive error surprises
Record Dates: First submitted 2024-03-22; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Refractive Errors
Keywords: refractive error surprises
MeSH Terms: conditions — Refractive Errors | interventions — Refractive Surgical Procedures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Corneal refractive surgery (Active Comparator): Among patients scheduled for cataract surgery, Group I; will undergo Corneal refractive surgery to correct any post-operative refractive surprises.
  Interventions: Procedure: Refractive surgeries
- IOL exchange (Active Comparator): Among patients scheduled for cataract surgery, Group II; will undergo IOL exchange to correct any post-operative refractive surprises.
  Interventions: Procedure: Refractive surgeries
- Piggyback sulcus IOL (Active Comparator): Among patients scheduled for cataract surgery, Group III; will undergo Piggyback sulcus IOL to correct any post-operative refractive surprises.
  Interventions: Procedure: Refractive surgeries

INTERVENTIONS:
Procedure: Refractive surgeries — after primary phacoemulsification surgery any resulting refractive error surprises will be corrected with different refractive surgery options

SUMMARY:
A refractive surprise can be defined as the failure to achieve the intended postoperative refractive target or the presentation of unexpected and, unwanted post-operative refractive error. It can cause anisometropia or dominance switch and is a source of patient dissatisfaction due to unmet expectations.The best way to manage refractive surprise is to prevent it. The 2017 NICE guidelines on the management of cataracts provide advice on prevention of refractive surprise through accurate biometry, A-constant optimisation, intraocular lens (IOL) formula selection and avoiding wrong lens implant errors.Benchmark standards for NHS cataract surgery dictate that 85% of eyes should be within 1 dioptre (D) and 55% within 0.5D of target spherical equivalent refraction following surgery.

DETAILED DESCRIPTION:
Aim(s) of the Research:

1. detection of refractive surprises using autorefractometer, and corneal topography.
2. treatment of the resulting refractive error surprises.

ELIGIBILITY:
Inclusion Criteria:

All adult patients scheduled for cataract surgery with:

* Symptomatizing patients with postoperative spherical error of more than 1 diopters.
* Symptomatizing patients with postoperative cylindrical error of more than 1 diopters.
* Symptomatizing patients with uncorrected distant visual acuity less than 6/24
* Symptomatizing patients with corrected distant visual acuity of less than 6/12
* Clear cornea. 6. Uneventful surgery.

Exclusion Criteria:

* Patients with complicated cataract.
* Raised intraocular pressure (IOP).
* Patients with pathologies of the posterior segment of the eye.
* Other causes of diminution of vision.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis and treatment of the resulting refractive error surprises | Baseline
  Rate of refractive error surprises

CONTACTS AND LOCATIONS:
Overall Officials: Magdy M Mostafa, MD, Study Director — Assiut University; Mohamed S Hussien, MD, Study Director — Assiut University; Ali N Ryad, MD, Study Director — Assiut University

REFERENCES:
- [Background] Abdelghany AA, Alio JL. Surgical options for correction of refractive error following cataract surgery. Eye Vis (Lond). 2014 Oct 16;1:2. doi: 10.1186/s40662-014-0002-2. eCollection 2014. PMID 26605349
- [Result] Day AC, Donachie PH, Sparrow JM, Johnston RL; Royal College of Ophthalmologists' National Ophthalmology Database. The Royal College of Ophthalmologists' National Ophthalmology Database study of cataract surgery: report 1, visual outcomes and complications. Eye (Lond). 2015 Apr;29(4):552-60. doi: 10.1038/eye.2015.3. Epub 2015 Feb 13. PMID 25679413
- [Result] Gale RP, Saldana M, Johnston RL, Zuberbuhler B, McKibbin M. Benchmark standards for refractive outcomes after NHS cataract surgery. Eye (Lond). 2009 Jan;23(1):149-52. doi: 10.1038/sj.eye.6702954. Epub 2007 Aug 24. PMID 17721503
- [Result] Khoramnia R, Auffarth G, Labuz G, Pettit G, Suryakumar R. Refractive Outcomes after Cataract Surgery. Diagnostics (Basel). 2022 Jan 19;12(2):243. doi: 10.3390/diagnostics12020243. PMID 35204334
- [Result] Moshirfar M, Thomson AC, Thomson RJ, Martheswaran T, McCabe SE. Refractive enhancements for residual refractive error after cataract surgery. Curr Opin Ophthalmol. 2021 Jan;32(1):54-61. doi: 10.1097/ICU.0000000000000717. PMID 33122488
- [Result] Ladas JG, Stark WJ. Improving cataract surgery refractive outcomes. Ophthalmology. 2011 Sep;118(9):1699-700. doi: 10.1016/j.ophtha.2011.05.038. No abstract available. PMID 21889661
- [Result] Iwase T, Tanaka N, Sugiyama K. Postoperative refraction changes in phacoemulsification cataract surgery with implantation of different types of intraocular lens. Eur J Ophthalmol. 2008 May-Jun;18(3):371-6. doi: 10.1177/112067210801800310. PMID 18465719